CLINICAL TRIAL: NCT04234633
Title: Effect of Gender on Clinical Presentation of SLE ِAt Assiut University Hospitals
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Safwat ِِِAbd elhamid eltaih, Principal Investigator, Assiut University
Other Study IDs: A44
Record Dates: First submitted 2020-01-11; First posted 2020-01-21 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: SLE

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SLE patients: Any SLE patients between 18 and 40 years old.

SUMMARY:
The investigators aim to compare the clinical characteristics and outcomes of SLE between male and female Egyptian patients at Assuit University Hospital.

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is an autoimmune disease of unknown etiology and is characterized by a multifaceted clinical presentation and disease course. Female predominance is a well-known characteristic of SLE, particularly during the reproductive years. Sex differences are another peculiarity of SLE with respect to clinical manifestations and outcomes. Previous studies have recognized male patients with lupus as a distinct minority; such patients often exhibit a poorer prognosis, especially involving the renal, cardiovascular, and neurologic systems. Higher mortality rates in male than in female patients with SLE have also been reported. Andrade et al reported that multiple conditions (for example, severe skin lesions, serositis, thrombotic events, and seizures) are more frequent in males than females.

Lu et al investigated the frequency of renal failure and end-stage renal disease among both genders and found out that these conditions were more prevalent among males. Another study shows no difference in complications and prognosis between both genders.

The results of these previous studies may not be applicable to all ethnic groups. For example, Mok et al studied the males in the local Chinese population had different disease features in term of clinical features at diagnosis, rate, and severity of relapse, organ damage and cumulative damage score. They found through a retrospective review that at the time of diagnosis, there was a trend, however not statistically significant, that males had less Raynaud's, alopecia, arthritis, anti-Ro antibody, but more thrombocytopenia and discoid lesions. Also, a significantly higher number of males had impaired renal functions.

There are few studies that have assessed the differences between male and female Egyptian patients with SLE according to the presentation, complication, prognosis, and mortality. One of these studies shows a more aggressive disease detected in male patients. This was evident by a higher prevalence of nephritis, fever, cutaneous vasculitis in male patients. on the other hand, alopecia and arthritis were significantly higher in females.

ELIGIBILITY:
Inclusion Criteria:

• Any SLE patients between 18and 40 years old will be eligible to be included in our study.

Exclusion Criteria:

* Patients below the age of 18 or above 40.
* Any other autoimmune disease.
* Cardiovascular, neurological, renal complications due to other co-morbidity such as DM and HTN.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Any SLE patients between 18and 40 years old will be eligible to be included in our study.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Presentation, complication, and mortality among males and female patients with SLE | 2 years
  Using percentages, we will track the number of patients that develop certain clinical conditions (such as arthritis, malar rash, .... ), complications (such as nephritis), and mortality rates. These numbers and percentages will be used to compare males with females (incidence rates for each event will be calculated).

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Aeltaih, MBBch, Principal Investigator — Assuit University Hospitals

IPD SHARING:
Plan to Share IPD: Undecided
No data will be shared.

REFERENCES:
- [Result] Mok CC, Lau CS, Chan TM, Wong RW. Clinical characteristics and outcome of southern Chinese males with systemic lupus erythematosus. Lupus. 1999;8(3):188-96. doi: 10.1191/096120399678847605. PMID 10342711
- [Result] Soto ME, Vallejo M, Guillen F, Simon JA, Arena E, Reyes PA. Gender impact in systemic lupus erythematosus. Clin Exp Rheumatol. 2004 Nov-Dec;22(6):713-21. PMID 15638045
- [Result] El Hadidi KT, Medhat BM, Abdel Baki NM, Abdel Kafy H, Abdelrahaman W, Yousri AY, Attia DH, Eissa M, El Dessouki D, Elgazzar I, Elgengehy FT, El Ghobashy N, El Hadary H, El Mardenly G, El Naggar H, El Nahas AM, El Refai RM, El Rwiny HA, Elsman RM, Galal M, Ghoniem S, Maged LA, Sally SM, Naji H, Saad S, Shaaban M, Sharaf M, Sobhy N, Soliman RM, El Hadidi TS. Characteristics of systemic lupus erythematosus in a sample of the Egyptian population: a retrospective cohort of 1109 patients from a single center. Lupus. 2018 May;27(6):1030-1038. doi: 10.1177/0961203317751856. Epub 2018 Feb 10. PMID 29431056